CLINICAL TRIAL: NCT03182764
Title: Policy-Related Survey - Territory-wide Telephone Survey on Tobacco Control
Brief Title: Tobacco Control-Related Policy Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Other Study IDs: 2017 Policy Survey
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Survey on Tobacco Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- never smokers: Never smokers are those who have never consumed cigarettes in their lifetime.
  Interventions: Other: No intervention
- Ex-smokers: Ex-smokers are those who consumed cigarettes previously but do not smoke at the time of the survey.
  Interventions: Other: No intervention
- Current smokers: Current smokers are those who, at the time of the survey, consume cigarettes daily or occasionally.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Aim: to collect further information on issues related to tobacco control which should be addressed and advocated in further tobacco control measures in Hong Kong

The objectives of this policy-related survey are as follows:

1. to update information on trends and prevalence of secondhand smoke, smoking attributable health effects, cessation services, and e-cigarette;
2. to investigate the level of public support on current and future tobacco control measures and taxation;
3. to address the timely impacts of smoke-free policies, public support for further tobacco control measures and assist COSH in shaping policy direction for government.

Current study is a cross-sectional retrospective telephone survey based on questionnaires. In total, 5,104 subjects will be randomly selected for a telephone interview. The subjects will be categorized into three groups, i.e. never smokers (1,700), ex-smokers (1,700) and current smokers (1,704). They will be required to answer a questionnaire via telephone. All data shall be collected using a Computer Assisted Telephone Interview (CATI) system, which allows real-time data capture and consolidation. All interviews shall be conducted anonymously. Analysis of survey data will aim to identify current opinion on tobacco control policies and implications for future policies. Analyses will be controlled for confounding variables as required by stratification into sub-groups based on important pre-defined characteristics and/or by multivariate analysis. Comparison with past trends and, where possible, extrapolation of future trends will be explored. Weights will be applied to adjust for the sex and age of Hong Kong population, and to handle the over-sampling issues of current smokers. The data analysis will be conducted by statisticians.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 or above
* Cantonese or Mandarin speakers

Exclusion Criteria:

* Unable to provide a consent form
* Speak language other than Cantonese and Mandarin

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Hong Kong residents
Sampling Method: Probability Sample
Enrollment: 5104 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-09-11 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Attitudes towards tobacco control policies | Finish all telephone survey by Sep 2017
  Topics included the awareness, use and perception of e-cigarettes, and public support for future tobacco control policies such as enlargement of graphic health warnings on cigarette packaging, tobacco tax increase and endgame.

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Public Opinion Programme, the University of Hong Kong, Hong Kong, Hong Kong